CLINICAL TRIAL: NCT03042091
Title: Combined Mechanical and Oral Antibiotic Bowel Preparation Versus Oral Antibiotics Alone for the Reduction of Surgical Site Infection Following Elective Colorectal Resection
Brief Title: Neomycin and Metronidazole Hydrochloride With or Without Polyethylene Glycol in Reducing Infection in Patients Undergoing Elective Colorectal Surgery
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16D.204
Record Dates: First submitted 2017-01-31; First posted 2017-02-03 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Colorectal Neoplasms; Diverticulitis; Inflammatory Bowel Diseases; Surgical Site Infection
MeSH Terms: conditions — Colorectal Neoplasms; Diverticulitis; Inflammatory Bowel Diseases; Surgical Wound Infection | interventions — Polyethylene Glycols; Ethanol; Glycols; polyethylene glycol 400; Neomycin; Metronidazole; Benchmarking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm I (mechanical bowel prep, oral antibiotics) (Active Comparator): Patients receive polyethylene glycol orally (PO), neomycin PO, and metronidazole hydrochloride PO on day -1. Patients undergo colorectal resection on day 0.
  Interventions: Drug: Polyethylene Glycol; Drug: Neomycin; Drug: Metronidazole Hydrochloride; Procedure: Therapeutic Conventional Surgery
- Arm II (oral antibiotics) (Experimental): Patients receive neomycin PO and metronidazole hydrochloride PO on day -1. Patients undergo colorectal resection on day 0.
  Interventions: Drug: Neomycin; Drug: Metronidazole Hydrochloride; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Polyethylene Glycol — Given orally
  Other Names: 25322-68-3; 57859; Ethanol; Glycol; Polyethylene Glycol 400
  Arms: Arm I (mechanical bowel prep, oral antibiotics)
Drug: Neomycin — Given orally
  Other Names: 1404-04-2; Neomycin Complex
Drug: Metronidazole Hydrochloride — Given orally
  Other Names: 69198-10-3; Flagyl; Metro I.V.; Satric
Procedure: Therapeutic Conventional Surgery — Undergo colorectal resection

SUMMARY:
This randomized clinical trial studies how well neomycin and metronidazole hydrochloride with or without polyethylene glycol work in reducing infection in patients undergoing elective colorectal surgery. Polyethylene glycol, may draw water from the body into the colon, flushing out the contents of the colon. Antibiotics, like neomycin and metronidazole hydrochloride, may stop bacteria from growing. It is not yet known whether it's better to give preoperative neomycin and metronidazole hydrochloride with or without polyethylene glycol in reducing surgical site infection after colorectal surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the difference in rates of surgical site infection following elective colorectal resections in patients given a preoperative mechanical bowel prep with oral antibiotics as compared to preoperative oral antibiotics alone.

SECONDARY OBJECTIVES:

I. To determine rates of post-operative clostridium difficile infection, adynamic ileus, cardiopulmonary complications, urinary tract infection, length of stay and mortality in patients given preoperative oral antibiotics with a mechanical bowel prep versus preoperative antibiotics alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing ileocolic resections, partial and total colectomies, and rectal resections for neoplasm, inflammatory bowel disease, or diverticulitis
* Subjects with the mental capacity to give informed consent

Exclusion Criteria:

* Patients undergoing emergent colorectal resections
* Patients who are decisionally-impaired and lack the mental capacity to give informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of post-operative surgical site infection (SSI) including superficial/incisional, deep, and organ space, anastomotic dehiscence and leak | Up to 30 days post operation
  The difference in incidence of SSI (antibiotics [ABX] - ABX + prep) will be calculated with an upper 95% confidence bound. Exploratory analysis will consider stratum specific estimates of differences in subgroups defined by BMI and diabetes status.

SECONDARY OUTCOMES:
Incidence of post-operative clostridium difficile infection | Up to 30 days post operation
  The difference in incidence of SSI (ABX - ABX + prep) will be calculated with an upper 95% confidence bound
Incidence of adynamic ileus | Up to 30 days post operation
  The difference in incidence of SSI (ABX - ABX + prep) will be calculated with an upper 95% confidence bound.
Incidence of cardiopulmonary complications | Up to 30 days post operation
  The difference in incidence of SSI (ABX - ABX + prep) will be calculated with an upper 95% confidence bound
Incidence of urinary tract infection | Up to 30 days post operation
  The difference in incidence of SSI (ABX - ABX + prep) will be calculated with an upper 95% confidence bound
Length of hospital stay | Up to 30 days post operation
Incidence of mortality | Up to 30 days post operation

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Phillips, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Willis MA, Toews I, Soltau SL, Kalff JC, Meerpohl JJ, Vilz TO. Preoperative combined mechanical and oral antibiotic bowel preparation for preventing complications in elective colorectal surgery. Cochrane Database Syst Rev. 2023 Feb 7;2(2):CD014909. doi: 10.1002/14651858.CD014909.pub2. PMID 36748942
- See also: Sidney Kimmel Cancer Center — http://www.kimmelcancercenter.org
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/